CLINICAL TRIAL: NCT03069807
Title: Can Latent Tuberculosis Infection (LTBI) in Recent Migrants be Treated Effectively and Safely in Primary Care? A Cluster Randomised Controlled Trial.
Brief Title: Completion and Acceptability of Treatment Across Primary Care and the commUnity for Latent Tuberculosis
Acronym: CATAPULT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: University College, London (Other); Public Health England (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 4212301
Record Dates: First submitted 2016-08-05; First posted 2017-03-03 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2018-01

CONDITIONS: Latent Tuberculosis
MeSH Terms: conditions — Latent Tuberculosis | interventions — Residence Characteristics; Primary Health Care

STUDY DESIGN:
Intervention Model Description: Cluster-randomised trial evaluating treatment completion (the primary outcome), uptake, acceptability, safety and cost-effectiveness of treating latent tuberculosis infection (LTBI) in migrants in primary care, compared with secondary care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants with LTBI will be treated in the Community/Primary Care.
  Interventions: Other: Community/Primary Care
- Control (Active Comparator): Participants with LTBI will be treated in the Hospital/TB Clinic
  Interventions: Other: Hospital/TB Clinic

INTERVENTIONS:
Other: Community/Primary Care — The treatment of Latent Tuberculosis Infection (LTBI) in the community by General Practitioners (Family Doctors) and Pharmacists
  Arms: Intervention
Other: Hospital/TB Clinic — The treatment of Latent Tuberculosis Infection (LTBI) in the Hospital TB Clinic by specialist doctors and nurses
  Arms: Control

SUMMARY:
This study investigates whether recent migrants to the United Kingdom are more likely to complete treatment for Latent Tuberculosis Infection (LTBI) if they are treated in the community (by General Practitioners/Family Doctors and pharmacists) than in a hospital TB clinic.

DETAILED DESCRIPTION:
People with dormant/latent TB (LTBI) have TB bacteria in their bodies, but do not have any symptoms because the bacteria are not active. The investigators know that recent migrants with LTBI from countries where TB is very common (incidence greater than 150 per 100 000) are at risk of developing active TB (their dormant bacteria become active) after they arrive in the UK. Active TB can be both infectious and deadly. The treatment for LTBI is three-month course of antibiotics. This significantly reduces the risk of developing active TB. This treatment is currently arranged and supervised by hospital clinics, however, many migrants do not attend and numbers of people completing antibiotics is low. This leaves many at risk of developing active TB. This study investigates whether a community (primary care) based approach to the treatment of LTBI, coordinated by general practices and local pharmacists, will achieve higher rates of antibiotic completion. The London Borough of Newham, in the UK, has amongst the highest rates of active TB in Western Europe. As part of a strategy to tackle this disease burden, an innovative model of care has been implemented in the borough in which GPs and pharmacists screen and treat migrants with LTBI. Our trial will evaluate whether primary care based management of LTBI leads to higher rates of treatment completion amongst recent migrants when compared to hospital based care. This approach would save money (both for the health service and for patients in terms of travels costs) and reduce numbers of new cases of active TB.

The treatment for Latent Tuberculosis Infection will be 3 months of combined oral Rifampicin and Isoniazid with Pyridoxine. The dosage is weight dependent.

ELIGIBILITY:
Inclusion Criteria:

* Patients with LTBI aged 16-35 and who have entered the UK less than 5 years ago from a country with a TB incidence of greater than 150/100,000.
* Latent Tuberculosis is defined as a positive IGRA test without any symptoms or physical signs of active Tuberculosis and no evidence of active Tuberculosis on Chest X-ray.

Exclusion Criteria:

1. Pregnant or breastfeeding women
2. Patients requiring medications that cannot be safely taken with Rifinah
3. HIV infection.
4. Individuals with known liver disease, or abnormal liver function tests (LFTs)
5. Diagnosis of cirrhosis (jaundice, haematemesis, ascites or previous episodes of liver encephalopathy)
6. Chronic or active hepatitis B or hepatitis C virus infection
7. Previous treatment for TB or LTBI.
8. Individuals who are unable to consent or who would usually be offered LTBI treatment under DOT because of their mental or social disabilities or those with drug or alcohol abuse
9. Evidence of active TB

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 362 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Completion of Latent Tuberculosis Treatment | 3 months
  Based on patients taking at least 90 percent of doses of Rifinah during 3 months of treatment.

SECONDARY OUTCOMES:
Complete of Latent Tuberculosis Treatment | 3 months
  Based on patients taking at least 80 or 85 percent of doses during 3 months of treatment.
Adherence to Treatment | 3 months
  To describe the proportion of individuals in the two treatment arms who adhere to LTBI treatment based on the five-point MARS5 (Medication Adherence Report Scale) questionairre, collection of prescriptions and a point of care urine testing for metabolites of isoniazid (Iso-screen) performed at monthly intervals.
Acceptability of Treatment | 3 months
  To describe the proportion of individuals in the two treatment arms who accept LTBI treatment. This is defined as those initiating treatment and attending TB clinics and community pharmacies on at least one occasion.
Adverse Effects of Treatment | 3 months
  To assess the incidence of adverse effects of treatment for LTBI, including adverse liver function tests or any other effects leading to cessation of treatment. This will be assessed using liver function test results, and a monthly questionnaire.
Active Tuberculosis | 2 years
  The incidence of active TB occurring within 2 years after enrolment. TB incidence in the intervention and control group will be compared and there will be a sub-analysis of examining those who did or did not accept or complete treatment. This will be performed through matching the study population with the national Enhanced TB Surveillance System, where information on all reported TB cases nationally are recorded.
Patient Satisfaction | 3 months
  Assessed using a standardised non-validated questionnaire (Likert scale)
Cost-effectiveness of Treatment | 2 years
  Assessed using a health economic model that includes locally and nationally agreed tariffs for latent tuberculosis treatment.
Patient Knowledge | 3 months
  The impact of patients knowledge about Latent Tuberculosis on treatment acceptance and completion will be assessed at baseline using a standardised non-validated questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Heinke Kunst, MD MSc, Principal Investigator — Queen Mary University of London
Locations (1):
- Shrewsbury Road Health Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Burman M, Zenner D, Copas AJ, Gosce L, Haghparast-Bidgoli H, White PJ, Hickson V, Greyson O, Trathen D, Ashcroft R, Martineau AR, Abubakar I, Griffiths CJ, Kunst H. Treatment of latent tuberculosis infection in migrants in primary care versus secondary care. Eur Respir J. 2024 Nov 7;64(5):2301733. doi: 10.1183/13993003.01733-2023. Print 2024 Nov. PMID 39174285
- [Derived] Burman M, Copas A, Zenner D, Hickson V, Gosce L, Trathen D, Ashcroft R, Martineau AR, Abubakar I, Griffiths C, Kunst H. Protocol for a cluster randomised control trial evaluating the efficacy and safety of treatment for latent tuberculosis infection in recent migrants within primary care: the CATAPuLT trial. BMC Public Health. 2019 Nov 29;19(1):1598. doi: 10.1186/s12889-019-7983-7. PMID 31783742